CLINICAL TRIAL: NCT06237270
Title: A Multicenter External Validation of a Novel Prediction Model for Elbow Flexion Recovery After Nerve Transfer Surgery in Brachial Plexus Injuries
Status: Completed | Type: Observational
Sponsor: Siriraj Hospital (Other)
Collaborators: Lerdsin General Hospital (Other)
Responsible Party: Principal Investigator, Panai Laohaprasitiporn, MD, Principal Investigator, Siriraj Hospital
Other Study IDs: 123/2566(IRB1), LH671009
Record Dates: First submitted 2024-01-23; First posted 2024-02-01 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2024-06

CONDITIONS: Brachial Plexus Injury
Keywords: nerve transfer; neurotization; brachial plexus injury; predictive factors; external validation; risk prediction model

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Successful biceps recovery: Motor power more than or equal to grade 3 at 24 months after surgery
  Interventions: Procedure: Nerve transfer surgery for elbow flexion
- Failure of biceps recovery: Motor power less than grade 3 at 24 months after surgery
  Interventions: Procedure: Nerve transfer surgery for elbow flexion

INTERVENTIONS:
Procedure: Nerve transfer surgery for elbow flexion — A functioning but less important nerve (e.g. spinal accessory nerve, phrenic nerve, fascicle of median nerve, or fascicle of ulnar nerve) was transferred to nerves innervating biceps or brachialis muscle to restore elbow flexion.

SUMMARY:
The goal of this observational study is to validate a risk prediction model developed for unsuccessful elbow flexion recovery after nerve transfer surgery in patients with brachial plexus injury. The main question it aims to answer is how well a risk prediction model perform in a different dataset, which are patients with brachial plexus injury who underwent surgery in a different time period or a different hospital.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic brachial plexus injury patients underwent nerve transfer operation for re-innervation of elbow flexion at Siriraj Hospital between 2018 and 2020 and Lerdsin General Hospital between 2008 and 2022
* Patients had follow-up duration at least 24 months after surgery

Exclusion Criteria:

* Incomplete medical records
* Patients underwent free functioning muscle transfer as primary surgery for elbow flexion
* Obstetric brachial plexus injury
* Radiation-induced brachial plexopathy

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Traumatic brachial plexus injury patients underwent nerve transfer operation
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-03-18 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with failure of biceps recovery at 24 months | 24 months
  Medical research council motor grading system of less than 3 at 24 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
Need a consensus from institute and colleagues